CLINICAL TRIAL: NCT04193241
Title: Suturing With U-technique Versus Un-Reapproximated Wound Edges During Removal of Closed Thoracostomy Tube Drain - A Single-centre Open-label Randomized Prospective Trial (SUTURE TRIAL)
Brief Title: Suturing With U-Technique Versus Un-Reapproximated Wound Edges During Removal of Closed Thoracostomy Tube Drain
Acronym: SUTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ibadan (Other)
Collaborators: Shalina Healthcare (Industry)
Responsible Party: Principal Investigator, Lateef Ayodele Baiyewu, MD, LECTURER/HONORARY CONSULTANT CARDIOTHORACIC SURGEON, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI/EC/18/0711; NHREC/05/01/2008a (Registry Identifier: UI/UCH ETHICS COMMITTEE)
Record Dates: First submitted 2019-11-29; First posted 2019-12-10 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pleural Effusion; Pneumothorax; Chest Trauma; Video-assisted Thoracoscopic Surgery; Thoracotomy; Pleural Diseases; Chylothorax; Empyema; Pyothorax; Thoracic Diseases; Thoracic Injury
Keywords: Chest tube insertion; Purse-string suture; occlusive adhesive-absorbent dressing; thoracostomy wound closure; wound complications; wound outcomes
MeSH Terms: conditions — Pleural Effusion; Pneumothorax; Thoracic Injuries; Pleural Diseases; Chylothorax; Empyema; Empyema, Pleural; Thoracic Diseases

STUDY DESIGN:
Intervention Model Description: 142 patients will be randomly assigned into two parallel groups of 71 each for each arm of the intervention
Masking Description: WinPepi software will be used to randomly assign the participants into either of the two arms of intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional purse-string suture closure (Active Comparator): A common-place conventional method of closure of chest tube or thoracostomy wound using a Prolene 1 purse-string suture (also known as U-suturing), at the time of chest tube removal.
  Interventions: Procedure: Closure of chest tube wound
- Suture-less occlusive-absorbent dressing closure (Experimental): Unconventional method of closing chest tube or thoracostomy wounds using Occlusive adhesive-absorbent dressing material (Primapore*) application i.e. Un-reapproximated wound edges, at time of chest tube removal
  Interventions: Procedure: Closure of chest tube wound

INTERVENTIONS:
Procedure: Closure of chest tube wound — At the time of chest tube removal, the chest tube site or thoracostomy wound will be closed in such a way as to prevent an iatrogenic pneumothorax or contamination of the pleural space
  Other Names: Thoracostomy wound closure

SUMMARY:
The study will be carried out by the principal investigator and his team at the Division of Cardiovascular and Thoracic Surgery of the Department of Surgery, College of Medicine, University of Ibadan and the University College Hospital, Ibadan (UCH), which is the Teaching Hospital of the Medical College.The study sets out to prospectively compare the early and long-term outcomes between the use of purse-string (suturing U-technique) and Un-reapproximated thoracostomy wound edges (Occlusive adhesive-absorbent dressing application) at the time of removal of thoracostomy tube drain in patients who have had chest tube insertion.

DETAILED DESCRIPTION:
Background: Closed thoracostomy tube drainage or chest tube insertion is one of the most commonly performed procedures in thoracic surgery. There are several published evidence-based guidelines on safe performance of a chest tube insertion. However, there is absence of any prospective controlled trial or systematic review, that scientifically proves the safest technique of closing the wound created at the time of chest tube insertion and that best guarantees good wound and overall outcomes, after chest tube removal. The use of a horizontal mattress non-absorbable suture or U- suture which is placed at the time of chest tube insertion and used to create a purse-string wound re-approximation at the time of tube removal, has been an age-long and time-honored practice in most thoracic surgical settings. It has been established by a fairly recent study that an occlusive adhesive-absorbent dressing can also be safely used to occlude the wound at the time of chest tube removal with good wound and overall outcomes though the study focused on tubes inserted during thoracic surgical operations.

Research Design: The study is an Open-label randomized prospective trial

Methodology: 142 consenting patients with indication for chest tube insertion, who meet the inclusion criteria for enrolment in the study will be randomly assigned into two balanced groups- Group A; that will have a Prolene 1 purse-string suture placed around the thoracostomy wound at the time of chest tube insertion and which will be used for the thoracostomy wound closure at the time of chest tube removal and Group B, that will not have a purse-string suture placement during chest tube insertion and will have their wounds covered by an occlusive adhesive-absorbent dressing material (Primapore*), at the time of chest tube removal. The procedure for chest tube insertion, indwelling chest tube management, post-tube removal care and outpatient follow-up; will be similar for both groups and will follow a pre-determined standardized protocol. Specific clinical outcomes while the chest tube is indwelling and specific clinical and wound outcomes after the chest tube removal will be observed in both Groups for comparison and to determine causal relationships. Observations will be recorded in a specially-designed study proforma.

ELIGIBILITY:
Inclusion Criteria:

Patients within the age limits who require chest tube insertion for any of the following indications:

1. Pleural effusion
2. Traumatic or spontaneous pneumothorax
3. Traumatic haemothorax
4. As an adjunct to a thoracotomy for a non-neoplastic and or non -infective condition

Exclusion Criteria:

Any patient so described above who has the following will be excluded:

1. An associated pyopneumothorax
2. Cancer encuirasse of the chest wall
3. Unconscious with unclear consent situation
4. With infective or neoplastic conditions of the chest wall
5. With individual or family history of wound failure e.g. unsightly scars
6. Who has had irradiation of the chest or chemotherapy administration within 6 weeks from the time of requirement of the chest tube insertion
7. Who is at risk of immunosuppression i.e. diabetes, HIV infection, on steroid therapy, ongoing chemotherapy or who has a congenital or any other acquired immune deficiency state
8. Presence of pleural adhesion during the process of chest tube insertion
9. Those with chest tube malposition after insertion, confirmed on chest radiograph, who will require tube adjustment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Proportion of clinical and wound complications with indwelling chest tube - SEVERE PAIN | It will span the period from chest tube insertion till chest tube removal
  Presence of severe pain at the chest tube site after chest tube insertion (Average daily pain score after tube insertion > 5 on the Visual Analog Scale and or Numerical Rating Scale)
Number of participants with clinical and wound complications with indwelling chest tube- TUBE DISLODGEMENT | It will span the period from chest tube insertion till chest tube removal
  Occurrence of tube dislodgement after chest tube insertion (expressed as "Present" or "Absent")
Number of participants with clinical and wound complications with indwelling chest tube - PERITUBAL LEAKAGE | It will span the period from chest tube insertion till chest tube removal
  Occurrence of peri-tubal leakage of fluid after chest tube insertion (expressed as "Present" or "Absent")
Number of participants with early wound complications after chest tube removal- AIR SUCK-IN | It will span the period from chest tube removal till the patient is discharged home after chest tube removal
  Presence of wound air suck-in after chest tube removal (indicated by presence of air suck-in sound through the wound into the pleural space during quiet and or forced inspiration)
Number of participants with early wound complications after chest tube removal- POST-INSERTION WOUND INFECTION | It will span the period from chest tube removal till the patient is discharged home after chest tube removal
  Occurrence of wound infection after chest tube removal (presence of purulent or offensive wound discharge with or without fever or presence of wound discharge that is microbiologically positive
Number of participants with early wound complications after chest tube removal- WOUND DEHISCENCE | It will span the period from chest tube removal till the patient is discharged home after chest tube removal
  Occurrence of wound dehiscence after chest tube removal (expressed as "Present" or "Absent")
Number of participants with early wound complications after chest tube removal- IATROGENIC PNEUMOTHORAX | It will span the period from chest tube removal till the patient is discharged home after chest tube removal
  Occurrence of early (within 7 days) and late pneumothorax (more than 1 week) after chest tube removal confirmed on chest radiography

SECONDARY OUTCOMES:
Number of participants with late wound complications after chest tube removal | After discharge from the hospital till 3 months after discharge
  Development of raised or elevated thoracostomy wound scars (unsightly scars appearing like hypertrophic scars or keloids) within 3 months of chest tube removal

CONTACTS AND LOCATIONS:
Overall Officials: Lateef A Baiyewu, MD,FWACS, Principal Investigator — College of Medicine University of Ibadan
Locations (1):
- Division of Cardiothoracic Surgery,Department of Surgery, University College Hospital,, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the trial, the study protocol, analytical plan and informed consent will be available for a 6 month window for asses by other researchers, reviewers or statutory institutions by email request or paper request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months
Access Criteria: By email request or paper request to the address of the Principal investigator as indicated above

REFERENCES:
- [Background] Martin M, Schall CT, Anderson C, Kopari N, Davis AT, Stevens P, Haan P, Kepros JP, Mosher BD. Results of a clinical practice algorithm for the management of thoracostomy tubes placed for traumatic mechanism. Springerplus. 2013 Dec 1;2:642. doi: 10.1186/2193-1801-2-642. eCollection 2013. PMID 24340246
- [Background] Monaghan SF, Swan KG. Tube thoracostomy: the struggle to the "standard of care". Ann Thorac Surg. 2008 Dec;86(6):2019-22. doi: 10.1016/j.athoracsur.2008.08.006. PMID 19022041
- [Background] Dural K, Gulbahar G, Kocer B, Sakinci U. A novel and safe technique in closed tube thoracostomy. J Cardiothorac Surg. 2010 Apr 6;5:21. doi: 10.1186/1749-8090-5-21. PMID 20370923
- [Background] Kim MS, Shin S, Kim HK, Choi YS, Kim J, Zo JI, Shim YM, Cho JH. Feasibility and Safety of a New Chest Drain Wound Closure Method with Knotless Sutures. Korean J Thorac Cardiovasc Surg. 2018 Aug;51(4):260-265. doi: 10.5090/kjtcs.2018.51.4.260. Epub 2018 Aug 5. PMID 30109204
- [Background] Yokoyama Y, Nakagomi T, Shikata D, Goto T. A novel technique for chest drain removal using a two layer method with triclosan-coated sutures. J Thorac Dis. 2017 Jan;9(1):211-213. doi: 10.21037/jtd.2017.01.31. PMID 28203426
- [Background] Chadwick AJ, Halfyard R, Ali M. Intercostal chest drains: Are you confident going on the pull? If not use the I-T-U approach. J Intensive Care Soc. 2015 Nov;16(4):312-325. doi: 10.1177/1751143715583856. Epub 2015 Apr 29. PMID 28979437
- [Background] Gilbert TB, McGrath BJ, Soberman M. Chest tubes: indications, placement, management, and complications. J Intensive Care Med. 1993 Feb-Mar;8(2):73-86. doi: 10.1177/088506669300800203. PMID 10148363
- [Background] Bertholet JW, Joosten JJ, Keemers-Gels ME, van den Wildenberg FJ, Barendregt WB. Chest tube management following pulmonary lobectomy: change of protocol results in fewer air leaks. Interact Cardiovasc Thorac Surg. 2011 Jan;12(1):28-31. doi: 10.1510/icvts.2010.248716. Epub 2010 Oct 6. PMID 20926462
- [Background] Vasseur BG. A simplified technique for closing thoracostomy incisions. Ann Thorac Surg. 2004 Apr;77(4):1467-8. doi: 10.1016/S0003-4975(03)01401-2. PMID 15063299
- [Background] Smelt JLC, Simon N, Veres L, Harrison-Phipps K, Bille A. The Requirement of Sutures to Close Intercostal Drains Site Wounds in Thoracic Surgery. Ann Thorac Surg. 2018 Feb;105(2):438-440. doi: 10.1016/j.athoracsur.2017.09.032. Epub 2017 Dec 7. PMID 29223423
- [Background] Rashid MA, Wikstrom T, Ortenwall P. A simple technique for anchoring chest tubes. Eur Respir J. 1998 Oct;12(4):958-9. doi: 10.1183/09031936.98.12040958. PMID 9817175
- [Background] Bosman A, de Jong MB, Debeij J, van den Broek PJ, Schipper IB. Systematic review and meta-analysis of antibiotic prophylaxis to prevent infections from chest drains in blunt and penetrating thoracic injuries. Br J Surg. 2012 Apr;99(4):506-13. doi: 10.1002/bjs.7744. Epub 2011 Dec 2. PMID 22139619
- [Background] Chan L, Reilly KM, Henderson C, Kahn F, Salluzzo RF. Complication rates of tube thoracostomy. Am J Emerg Med. 1997 Jul;15(4):368-70. doi: 10.1016/s0735-6757(97)90127-3. PMID 9217527
- [Background] Helling TS, Gyles NR 3rd, Eisenstein CL, Soracco CA. Complications following blunt and penetrating injuries in 216 victims of chest trauma requiring tube thoracostomy. J Trauma. 1989 Oct;29(10):1367-70. doi: 10.1097/00005373-198910000-00013. PMID 2810412
- [Background] Walming S, Angenete E, Block M, Bock D, Gessler B, Haglind E. Retrospective review of risk factors for surgical wound dehiscence and incisional hernia. BMC Surg. 2017 Feb 22;17(1):19. doi: 10.1186/s12893-017-0207-0. PMID 28222776
- [Background] Singer AJ, Hollander JE, Quinn JV. Evaluation and management of traumatic lacerations. N Engl J Med. 1997 Oct 16;337(16):1142-8. doi: 10.1056/NEJM199710163371607. No abstract available. PMID 9329936
- [Background] Yag-Howard C. Sutures, needles, and tissue adhesives: a review for dermatologic surgery. Dermatol Surg. 2014 Sep;40 Suppl 9:S3-S15. doi: 10.1097/01.DSS.0000452738.23278.2d. PMID 25158874
- [Background] Burkhardt R, Lang NP. Influence of suturing on wound healing. Periodontol 2000. 2015 Jun;68(1):270-81. doi: 10.1111/prd.12078. PMID 25867989
- [Background] Sonmez K, Bahar B, Karabulut R, Gulbahar O, Poyraz A, Turkyilmaz Z, Sancak B, Basaklar AC. Effects of different suture materials on wound healing and infection in subcutaneous closure techniques. B-ENT. 2009;5(3):149-52. PMID 19902850
- [Background] Mirkovic S, Selakovic S, Sarcev I, Bajkin B. Influence of surgical sutures on wound healing. Med Pregl. 2010 Jan-Feb;63(1-2):7-14. doi: 10.2298/mpns1002007m. English, Serbian. PMID 20873303
- [Background] Scheidel P, Hohl MK. Modern synthetic suture materials and abdominal wound closure techniques in gynaecological surgery. Baillieres Clin Obstet Gynaecol. 1987 Jun;1(2):223-46. doi: 10.1016/s0950-3552(87)80052-4. PMID 2961498
- [Background] Gazivoda D, Pelemis D, Vujaskovic G. A clinical study on the influence of suturing material on oral wound healing. Vojnosanit Pregl. 2015 Sep;72(9):765-9. doi: 10.2298/vsp140401064g. PMID 26554107
- [Background] Zeplin PH, Schmidt K, Laske M, Ziegler UE. Comparison of various methods and materials for treatment of skin laceration by a 3-dimensional measuring technique in a pig experiment. Ann Plast Surg. 2007 May;58(5):566-72. doi: 10.1097/01.sap.0000245135.58229.e7. PMID 17452845
- [Background] Tejani C, Sivitz AB, Rosen MD, Nakanishi AK, Flood RG, Clott MA, Saccone PG, Luck RP. A comparison of cosmetic outcomes of lacerations on the extremities and trunk using absorbable versus nonabsorbable sutures. Acad Emerg Med. 2014 Jun;21(6):637-43. doi: 10.1111/acem.12387. PMID 25039547
- [Background] Helfman T, Ovington L, Falanga V. Occlusive dressings and wound healing. Clin Dermatol. 1994 Jan-Mar;12(1):121-7. doi: 10.1016/0738-081x(94)90262-3. No abstract available. PMID 8180934
- [Background] Rovee DT. Evolution of wound dressings and their effects on the healing process. Clin Mater. 1991;8(3-4):183-8. doi: 10.1016/0267-6605(91)90030-j. PMID 10149169
- [Background] Kannon GA, Garrett AB. Moist wound healing with occlusive dressings. A clinical review. Dermatol Surg. 1995 Jul;21(7):583-90. doi: 10.1111/j.1524-4725.1995.tb00511.x. PMID 7606367
- [Background] Hutchinson JJ, Lawrence JC. Wound infection under occlusive dressings. J Hosp Infect. 1991 Feb;17(2):83-94. doi: 10.1016/0195-6701(91)90172-5. PMID 1674265
- [Background] Triller C, Huljev D, Planinsek Rucigaj T. [Modern wound dressings]. Acta Med Croatica. 2013 Oct;67 Suppl 1:81-7. Croatian. PMID 24371980
- [Background] Abramson JH. WINPEPI updated: computer programs for epidemiologists, and their teaching potential. Epidemiol Perspect Innov. 2011 Feb 2;8(1):1. doi: 10.1186/1742-5573-8-1. PMID 21288353
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT04193241/Prot_SAP_ICF_000.pdf